CLINICAL TRIAL: NCT00181922
Title: Open-Label Study of Ziprasidone for the Treatment of Mania in Children and Adolescents With Bipolar Spectrum Disorder
Brief Title: Ziprasidone for the Treatment of Mania in Children and Adolescents With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002-p-000183
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar Disorder; Mania
Keywords: bipolar disorder; children; ziprasidone; mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — ziprasidone

INTERVENTIONS:
Drug: ziprasidone (Geodon)

SUMMARY:
The objective of this study is to compare the safety and effectiveness of Ziprasidone in the treatment of mania in children and adolescents with Bipolar disorder over 8 weeks. This is an exploratory, open-label study, which seeks to determine if there is evidence for efficacy. The results of this study will be used to generate hypotheses for a larger study.

DETAILED DESCRIPTION:
Initial clinical evidence suggests that atypical neuroleptics may play a unique therapeutic role in the management of symptoms in youth with bipolar disorder. Ziprasidone is classed as an atypical neuroleptic because of its unique pharmacological profile that includes both D2 and 5HT2 antagonistic effects. This combined dopaminergic and serotonergic activity seems to be associated not only with antipsychotic effects but also with mood stabilizing, mood elevating and anti-aggressive effects as well as a lower risk for extrapyramidal symptoms and tardive dyskinesia.

Ziprasidone in particular has been found to have a higher 5HT2A to D2 receptor affinity ratio, which suggests that the likelihood of extrapyramidal symptoms and hyperprolactinemia may be further decreased. This makes it an ideal candidate to treat mania in children, but although it is used in clinical practice, adequate data has not been collected on its safety and effectiveness. This study included 1) an 8-week acute period, during which participants were observed during weekly visits, and up to a 10-month extension period, during which participants saw a study clinician on a monthly basis, to document the response rate 2) assessment of the impact of Ziprasidone on functional capacities (quality of life, psychosocial function) and cognition, 3) careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 6 to 18 years of age
2. Parent or legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
3. Patients and their legal representative must be considered reliable.
4. Each patient and his/her authorized legal representative must understand the nature of the study. The patient's authorized legal representative must sign an informed consent document.
5. Patient must have a diagnosis of bipolar I or bipolar II disorder and currently displaying an acute manic, hypomanic, or mixed episode (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders).
6. Patients must have an initial score on the Y-MRS total score of at least 15.
7. Patient must be able to participate in mandatory blood draws.
8. Patient must be able to swallow pills.

Exclusion Criteria:

1. Patients with chronic medical illness, DSM-IV substance dependence within the past 6 months, pregnant or nursing females, and those at serious risk of suicide will be excluded from the study
2. investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
3. Serious unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
4. Known history of QT prolongation (ie. Congenital long QT syndrome), cardiac arrhythmia, recent myocardial infarction, or heart failure
5. Concurrent medications known to prolong the QT interval including: antiarrhythmics (quinidine), antimicrobials and antimalarials (erythromycin, clarithromycin, ketoconazole, sparfloxacin, moxifloxacin, levofloxacin, gatifloxacin, chloroquine) and antihistamines (diphenhydramine, hydroxyzine).
6. Known hypokalemia or hypomagnesemia
7. Uncorrected hypothyroidism or hyperthyroidism
8. History of severe allergies or multiple adverse drug reactions
9. Non-febrile seizures without a clear and resolved etiology
10. Leukopenia or history of leucopenia without a clear and resolved etiology
11. DSM-IV substance (except nicotine or caffeine) dependence within the past 6 months
12. Judged clinically to be at serious suicidal risk
13. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol
14. History of intolerance of Ziprasidone as determined by the principal investigator.
15. Treatment with an irreversible monoamine oxidase inhibitor within 2 weeks prior to visit 2
16. Current diagnosis of schizophrenia
17. For concomitant stimulant therapy used to treat ADHD, patients must have been on a stable dose of medication for 1 month prior to randomization

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2002-03; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
reduction in symptoms assessed by
Clinical Global Improvement scale (Severity, Improvement and Efficacy Index)
Young Mania Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Cambridge, Massachusetts